CLINICAL TRIAL: NCT05639543
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Dose-Escalation, Proof-of-Concept Study Evaluating the Safety, Tolerability, Efficacy and Pharmacokinetics of INT-787 in Subjects With Severe Alcohol Associated Hepatitis
Brief Title: FXR Effect on Severe Alcohol-Associated Hepatitis (FRESH) Study
Acronym: FRESH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 787-201
Record Dates: First submitted 2022-11-09; First posted 2022-12-06 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Associated Hepatitis
Keywords: Severe Alcohol associated Hepatitis (sAH); Alcoholic Hepatitis (AH); Hepatitis; Alcoholic
MeSH Terms: conditions — Hepatitis, Alcoholic; Hepatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- INT-787 (Active Comparator): Participants will be randomized to receive INT-787 (in Dose Escalation Cohorts [Cohorts 1 through 4] and Extension Phase Cohorts [Cohorts 5 and 6])
  Interventions: Drug: INT-787
- Placebo (Placebo Comparator): Participants will be randomized to receive matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INT-787 — Blinded Study Drug
  Arms: INT-787
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this trial is to assess dose related safety, efficacy, and pharmacokinetics (PK) of INT-787 in participants with severe alcohol-associated hepatitis (sAH).

DETAILED DESCRIPTION:
This is a Phase 2a, randomized, double-blind, placebo-controlled, dose-escalation, proof-of-concept study to evaluate the safety, tolerability, efficacy, and PK of INT-787 in participants, initially admitted to the hospital, with severe alcohol-associated hepatitis (sAH). The study aims to demonstrate and provide rationale for the selection of optimal dose(s) of INT-787 in the target population of participants with sAH. INT-787 will be evaluated for safety and tolerability prior to dose escalation. Overall efficacy, compared to placebo, will be assessed for each dose cohort.

Additionally, PK measurements at various study timepoints will allow the Sponsor to better understand the systemic exposure of INT-787 and the relationship between exposure and efficacy and safety. Such insights in participants with more advanced liver disease will provide valuable information for future clinical trials of INT-787.

The placebo-treated participants will provide important natural history information on outcomes in this participant population with sAH treated with supportive care. The placebo-treated participants within cohorts are meant to blind the study drug administration while the data across dose cohorts will be used in the overall analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 to 65 years (inclusive)
2. Clinical diagnosis of sAH based on all the following:

   1. History of ongoing excess alcohol (>60 g/day [male] or >40 g/day [female]) use for ≥6 months, with <60 days of abstinence prior to the onset of jaundice
   2. Serum total bilirubin >3.0 mg/dL
   3. Aspartate aminotransferase (AST) ≥50 U/L
   4. AST/Aspartate aminotransferase (ALT) ratio ≥1.5
   5. Onset of jaundice within prior 8 weeks
   6. Cohort 1 through Cohort 4: Maddrey's Discriminant Factor (mDF) ≥32 and ≤70
   7. Cohort 5 and Cohort 6: mDF ≥32
3. Cohort 1 through Cohort 4: MELD score ≥18 to ≤25 (inclusive) and Cohort 5 and Cohort 6: MELD score ≥21 to ≤30
4. Female participants must be postmenopausal, surgically sterile, or, if premenopausal (and not surgically sterile), be prepared to use ≥1 highly effective method of contraception from the initiation of Screening and for 90 days after the last dose of investigational product as follows:

   * Surgical sterilization (bilateral tubal occlusion, etc.)
   * Placement of an intrauterine device (IUD) or intrauterine system (e.g., intrauterine hormone-releasing system [IUS])
   * Combined (estrogen and progesterone containing) hormonal contraceptive associated with inhibition of ovulation:

     * Oral
     * Intravaginal
     * Transdermal
   * Progesterone-only hormonal contraception associated with inhibition of ovulation:

     * Oral
     * Injectable
     * Implantable
   * Sexual abstinence: When in line with the preferred and usual lifestyle of the participant, is defined as avoiding all types of activity that could result in conception (pregnancy) from the initiation of Screening and until at least 90 days after the last dose of investigational product
5. Male participants who are sexually active with female partners of childbearing potential must agree to use a condom with spermicide and to use 1 other approved method of highly effective contraception from the initiation of Screening and until at least 90 days after the dose of investigational product as listed in Inclusion Criteria #3.
6. Male participants must refrain from sperm donation from the initiation of Screening and until at least 90 days after the last dose of investigational product
7. Must provide written informed consent and agree to comply with the study protocol. In participants with hepatic encephalopathy which may impair decision-making, consent will be obtained per hospital procedures (e.g., by Legally Authorized Representative).
8. Participants must agree to participate in an alcohol use disorder program during the study period, as recommended by the local institution's addiction medicine specialists, including post-hospitalization

Exclusion Criteria:

1. Participants taking products containing obeticholic acid in the 30 days prior to randomization
2. Participants taking >2 doses of systemic corticosteroids within 30 days prior to randomization.
3. Participants who have been inpatient at a referral hospital for >7 days prior to transfer.
4. Pregnancy, planned pregnancy, potential for pregnancy (e.g., unwillingness to use effective birth control during the study), or current or planned breast feeding.
5. Abstinence from alcohol consumption for >2 months before Day 1.
6. AST or ALT >400 U/L.
7. Cohort 1 through Cohort 4: mDF <32 or >70.
8. Cohort 5 and Cohort 6: mDF <32
9. Cohort 1 through Cohort 4: MELD score <18 or >25.
10. Cohort 5 and Cohort 6: MELD <21 or >30
11. Other causes of liver disease including chronic hepatitis B (hepatitis B surface antigen [HBsAg] positive), chronic hepatitis C virus (HCV) RNA positive, drug-induced liver injury (DILI), biliary obstruction, and autoimmune liver disease.
12. Current or previous history of hepatocellular carcinoma (HCC)
13. History of liver transplantation or currently listed for liver transplant
14. Untreated infection (e.g., has not initiated appropriate medical treatment for infection)
15. Known positivity for human immunodeficiency virus infection
16. Uncontrolled gastrointestinal (GI) bleeding or controlled GI bleeding that was associated with shock or required transfusion of more than 3 units of blood within 7 days of Screening.
17. Kidney injury defined as a serum creatinine >133 μmol/L (>1.5 mg/dL) or the requirement for renal replacement therapy whether prior to or after study screening.
18. Portal vein thrombosis
19. Acute pancreatitis or acute gallbladder disease (e.g., cholecystitis)
20. Severe, on-going associated disease (e.g., cardiac failure, acute myocardial infarction, severe cardiac arrhythmias, severe pulmonary disease, neurologic disease)
21. Malignancy within the 2 years prior to Screening, with the exception of specific cancers that have been cured by surgical resection (e.g., basal cell skin cancer). Participants under evaluation for possible malignancy are not eligible.
22. Positive urine drug screen (amphetamines, barbiturates, benzodiazepines, cocaine, and opiates) except tetrahydrocannabinol or in the setting of documented prescription medications (e.g., opiates, benzodiazepines, amphetamines, barbiturates), which also include medications prescribed as part of in-patient management. Participants being treated for alcohol withdrawal may be exempt for this reason, verify with Medical Monitor.
23. Participated in a clinical research study and received any active investigational product being evaluated for the treatment of sAH within 3 months before Day 1
24. Participation in a study of another investigational medicine or device within 30 days before Screening
25. Any other condition or clinical laboratory result that, in the opinion of the Investigator, might confound the results, or would impede compliance or hinder completion of the study
26. Participants treated in the Dose Escalation Phase (Cohort 1 through Cohort 4) are not eligible for enrollment into an Extension Cohort (Cohort 5 and Cohort 6), and participants treated in Cohort 5 are not eligible for enrollment into Cohort 6.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2026-09-06 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Lille model response based on Lille score by treatment group | Day 7
  The Lille score response rate will be analyzed as a categorical variable. Participants with Lille score <0.45 will be counted as responders and those with Lille score ≥0.45 will be counted as non-responders.

SECONDARY OUTCOMES:
Change from baseline in the Model for End-Stage Liver Disease (MELD) score at 28-days by treatment group | Baseline and at Day 28
  The MELD scoring system is used to assess the severity of liver disease in participants in the setting of alcohol-associated hepatitis. The MELD score is derived from the participant's serum total bilirubin, serum creatinine, and international normalized ratio (INR). The MELD score ranges from 6 to 40 with higher scores indicating more severe liver disease and a worse outcome.
Change from Baseline in total bilirubin | Baseline and at Day 7, 14, 21, 28, 56 and 84
Difference in 28-day, 56-day, and 84-day all-cause mortality or liver transplantation (TFS) between INT-787 and placebo | Day 28, 56, 84
Number of participants with treatment emergent adverse events (TEAEs), serious adverse events (SAEs) and treatment emergent adverse event of special interest (AESIs) | During the study period, up to 12 weeks
Number of participants reporting infectious adverse events by System organ class (SOC)/ preferred term by treatment group | During the study period, up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (31):
- United States (21):
  - Stanford Healthcare, Palo Alto, California
  - Clinical Translational Research Site, Miami, Florida
  - Tampa General Medical Group, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Mercy Medical Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Rutgers-New Jersey Medical School, Newark, New Jersey
  - Northwell Health Center for Liver Disease and Transplantation, Manhasset, New York
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt Digestive Disease Center, Nashville, Tennessee
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Parkland Health and Hospital System, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - VCU Health Clinical Research Services Unit, Richmond, Virginia
- France (5):
  - CHU Angers, Angers, France
  - Hopital Beaujon, Clichy
  - Hopital Claude Huriez, Lille
  - Hopital Pitie Salpetriere, Paris
  - Hopital Rangueil, Toulouse
- United Kingdom (5):
  - Cambridge University NHS Foundation Trust, Cambridge
  - Royal Free Hospital, London
  - Imperial College Healthcare NHS Trust, London
  - King's College Hospital, London
  - University Hospitals Plymouth NHS Trust, Plymouth

IPD SHARING:
Plan to Share IPD: No